CLINICAL TRIAL: NCT01508780
Title: Combined Use of Angiography, Optical Coherence Tomography and Intravascular Ultrasound in Evaluation of Pulmonary Vascular Structure and Function in Patients With Pulmonary Arterial Hypertension Treated With Oral Bosentan
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to complex study protocol, no patients have been enrolled in the study.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011P000916
Record Dates: First submitted 2012-01-03; First posted 2012-01-12 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

ARMS (1):
- Pulmonary Arterial Hypertension, bosentan (Experimental): Subjects include patients being diagnosed with pulmonary arterial hypertension and starting treatment with bosentan.
  Interventions: Device: St Jude Medical C7 Dragonfly Optical Coherence Tomography (OCT); Device: Boston Scientific Intravascular Ultrasound

INTERVENTIONS:
Device: St Jude Medical C7 Dragonfly Optical Coherence Tomography (OCT) — All subjects will have OCT and IVUS imaging during their right heart catheterization.
Device: Boston Scientific Intravascular Ultrasound — All subjects will have OCT and IVUS imaging during their right heart catheterization.

SUMMARY:
It has been hypothesized that one of the benefits of bosentan relates to pulmonary vascular remodeling. The investigators believe that this study will help document the nature of beneficial changes that occur in patients with Pulmonary Arterial Hypertension (PAH) in response to bosentan therapy. In turn, demonstrating that changes in pulmonary vascular structure and function accompany clinical improvement.

DETAILED DESCRIPTION:
Subjects will have Optical coherence tomography (OCT) and Intravascular Ultrasound (IVUS) imaging during the right heart catheterization that diagnoses them as having PAH. Subjects will start their bosentan and will be followed by monthly clinic visits for 4 months. At 4 months they will have repeat OCT and IVUS imaging.

ELIGIBILITY:
Inclusion Criteria:

1. WHO GROUP 1
2. AGE 18-75
3. Baseline 6-min walk distance (6MWD) between 200 and 450 m
4. Diagnosed with pulmonary artery hypertension during right heart catheterization (Mean Pulmonary Artery Pressure > 25mmHg)

General Exclusion Criteria

1. Pregnant or nursing
2. Acute or chronic illness other than those associated with PAH (collagen vascular disease, human immunodeficiency virus, or anorexigen use)
3. Previously received any investigational medications, prostanoids, or phosphodiesterase inhibitors
4. eGFR < 60
5. Angina
6. Syncope
7. Failing right ventricle
8. Hemoptysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in the measurement of Pulmonary arterial intimal + Medial thickening by OCT pre and post treatment with bosentan at 4 months | Baseline and 4 months

SECONDARY OUTCOMES:
Change in pulmonary arterial pulsatility by IVUS pre and post treatment with bosentan at 4 months | Baseline and 4 months
Change in pulmonary arterial pressure/elastic strain index by IVUS pre and post treatment with bosentan at 4 months | Baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States